CLINICAL TRIAL: NCT04390425
Title: Limb Occlusion Pressure Tourniquets to Decrease Pain After Surgery
Acronym: LOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shari Liberman, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00018544
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Limb Occlusion Pressure

STUDY DESIGN:
Intervention Model Description: There are two groups for this study. The control group receives standard pneumatic tourniquet pressure and the experimental group receives limb occlusion pressure. It is randomized and double-blinded.
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor the operating surgeon know the which group the subject is randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control - Standard pneumatic tourniquet pressure (No Intervention): This group receives the standard pneumatic tourniquet pressure during surgery like they would during standard of care.
- Experimental - Limb occlusion pressure (Experimental): This group receives a slightly lower tourniquet pressure than they would during standard of care. This lowered limb occlusion pressure is determined by the tourniquet device.
  Interventions: Device: Experimental - Limb Occlusion pressure

INTERVENTIONS:
Device: Experimental - Limb Occlusion pressure — This intervention involves lower tourniquet pressure than the standard of care. There is no change to tourniquet time or how the surgery is performed.
  Arms: Experimental - Limb occlusion pressure

SUMMARY:
Currently a standard tourniquet pressure is used for orthopedic surgeries. High tourniquet pressure had been associated with adverse side effects such as ischemia, muscle weakness, and post operative pain. Limb Occlusion Pressure, LOP, is based off the patient's systolic blood pressure plus a safety margin and is typically much lower than standard tourniquet pressure. The aim of this study is to determine if using LOP during orthopedic surgeries decreases post-operative pain and opioid consumption and improves patient's outcomes.

DETAILED DESCRIPTION:
The study will start for each subject in the clinic setting during a standard pre-operative office visit. Consent for the study will be obtained after explaining all aspects of the study. The subjects will be randomly separated into two groups. Half of the subjects will have their procedure performed under standard tourniquet pressure, and the other half of the subjects will have their procedure performed with a distal photoplenthysmography probe that will calculate Limb Occlusion Pressure and inflate the tourniquet to the calculated Limb Occlusion Pressure. The subject will undergo their scheduled procedure in the operating room. The subject will also keep a daily pain and opioid consumption diary at home for two weeks after the surgery. The subject will complete patient outcome questionnaires before the surgery, two weeks after the operation, and 8 weeks after the operation to assess patient outcomes. The subject can complete the questionnaires at home, but if they do not, they will have the option to fill the out during their clinic visits. The patient's pre and post OP questionaries' will be the indicators for patient outcomes. All of the standardized questionnaires give calculated scores based off the patients' responses. As the subject improves their score will increase.The research team can compare change in score between the two groups and change with in groups to access patient outcomes.

To maintain the double blind nature of the study, the tourniquet will be placed, inflated, and draped over before the surgeon enters the operating room. Someone else on the research team, one of the coordinators or one of the residents will record the patients' systolic blood pressure and cuff pressure of the tourniquet before the attending enters the OR. This way the surgeon is still blind to the cuff pressure technique used, LOP or STP, when they rate the quality of the bloodless field after the surgery using a VAS scale.

All of these documents are attached on the summary page under additional documents on the Psycho-Physiological Testing page under number 1. List all the measures/instruments that will be used for this study. The VAS pain and opioid consumption diary is titled LOP pain diary cover page and LOP pain diary. The questionnaires that will be used are DASH, IKDC Subject Knee Evaluation Form, KOOS Junior, KOOS Lysholm, Marx, Michigan Hand Outcomes, Patient Rated Wrist Evaluation, Promis Bank v 1.2 Physical Function, PROMIS SF v 1.1 Global Health, and Tegner Activity Level Scale.

ELIGIBILITY:
Inclusion Criteria:

* The research team will test the central hypothesis that LOP tourniquets will decrease pain and opioid use and improve patients outcomes on healthy adults (above the age of 18) undergoing either open carpal tunnel release, open reduction internal fixation distal radius fracture, cubital tunnel release, trigger finger release, thumb CMC arthroplasty, anterior cruciate ligament reconstruction, or total knee replacements

Exclusion Criteria:

1. Prescription pain medications for chronic conditions (> 6 weeks)
2. Patients who cannot use a tourniquet:( ex. Certain patients with fistulas or PVD, certain patient with Peripheral Vascular Disease)
3. Prior trauma or surgery to the observed limb.
4. Hypotension or hypertension that prevents accurate distal photoplenthysmography probe reading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative surgical site pain | Pain will be recorded as an average of three reported VAS recordings throughout each day for 14-days following surgery. Will compare change in average pain relative baseline pre-op (0) (within group) at each day post-surgery for 14 days
  Visual analog scale from 0 (no pain) to 10 (worst pain imaginable)
Postoperative tourniquet site pain | Pain will be recorded as an average of three reported VAS recordings throughout each day for 14-days following surgery. Will compare change in average pain relative baseline pre-op (0) (within group) at each day post-surgery for 14 days
  Visual analog scale from 0 (no pain) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Postoperative opioid usage | Once a day, every day for 2 weeks postoperatively
  Patients record the name of the opioid, dosage, and number of pills taken. These are standardized using the morphine milligram equivalents formula.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aflatooni J, Goble H, Lambert B, Liberman S, McCulloch PC. Limb Occlusion Pressure Versus Standard Pneumatic Tourniquet Pressure in Anterior Cruciate Ligament Surgery: A Randomized Controlled Trial. J Am Acad Orthop Surg Glob Res Rev. 2025 Apr 30;9(5):e24.00282. doi: 10.5435/JAAOSGlobal-D-24-00282. eCollection 2025 May 1. PMID 40326965